CLINICAL TRIAL: NCT02644668
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Multiple Dose Study of CK-2127107 in Two Ascending Dose Cohorts of Patients With Spinal Muscular Atrophy
Brief Title: A Study of CK-2127107 in Patients With Spinal Muscular Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CY 5021
Record Dates: First submitted 2015-12-23; First posted 2016-01-01 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Spinal Muscular Atrophy
Keywords: Reldesemtiv
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — reldesemtiv

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Patients randomized to this treatment arm will receive a placebo suspension twice daily for 8 weeks.
  Interventions: Drug: Placebo
- Reldesemtiv 150 mg twice daily (Experimental): Patient randomized to this treatment arm will receive reldesemtiv suspension at a dose of 150 mg, twice daily for 8 weeks.
  Interventions: Drug: Reldesemtiv 150 mg
- Reldesemtiv 450 mg twice daily (Experimental): Patients randomized to this treatment arm will receive reldesemtiv suspension at a dose of 450 mg, twice daily for 8 weeks.
  Interventions: Drug: Reldesemtiv 450 mg

INTERVENTIONS:
Drug: Placebo — Granules for oral suspension (placebo)
  Arms: Placebo
Drug: Reldesemtiv 150 mg — Granules for oral suspension, 18.7% reldesemtiv
  Other Names: CK-2127107
  Arms: Reldesemtiv 150 mg twice daily
Drug: Reldesemtiv 450 mg — Granules for oral suspension, 56.0% reldesemtiv
  Other Names: CK-2127107
  Arms: Reldesemtiv 450 mg twice daily

SUMMARY:
This study will evaluate the pharmacodynamic (PD) effect of CK-2127107 (hereafter referred to as reldesemtiv) versus placebo on measures of skeletal muscle function or fatigability in patients with Type II, III, or IV spinal muscular atrophy (SMA).

DETAILED DESCRIPTION:
CY 5021 is a Phase 2, double-blind, randomized, placebo-controlled, multiple dose study of reldesemtiv in 2 sequential ascending dose cohorts of patients with SMA. Patients will be randomized 2:1 to receive reldesemtiv or placebo twice daily for 8 weeks. Patients randomized to reldesemtiv in Cohort 1 will receive a dose of 150 mg twice daily and patients randomized to reldesemtiv in Cohort 2 will receive 450 mg twice daily. Within each cohort, randomization will be stratified by ambulatory status (ambulatory versus non ambulatory).

The primary objective of the study is to determine the PD effects of reldesemtiv on measures of pulmonary function, respiratory function, muscle strength, and motor function. Other PD measures include changes in the timed up and go (TUG) test, a 6-minute walk test (6MWT), and patient and investigator global assessments. Secondary objectives include the safety of multiple doses of reldesemtiv and an evaluation of the pharmacokinetics of reldesemtiv.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an Informed Consent Form (ICF) for patients 18 years of age and older. For patients less than 18 years of age, parent(s)/legal guardian(s) of patients must provide written informed consent prior to participation in the study and informed assent will be obtained from minors at least 12 years of age when required by regulation.
* Males or females with genetically confirmed diagnosis of SMA who are Type II, III or IV and at least 12 years of age
* Ambulatory patients, once having achieved a standing position independently, must be able to complete at least one lap in the 6-minute walk test (at least 50 meters) within 6 minutes without assistance.
* Non-ambulatory patients (defined as individuals who are effectively requiring a wheelchair for all mobility needs; they may be able to stand or walk short distances, but unable to walk 50 meters without assistance in 6 minutes). Non-ambulatory patients must be able to tolerate an upright sitting position, with support, continuously for 3 hours
* Hammersmith (HFMS-E) score ≥ 10 and ≤ 54
* Contracture of the elbow flexion and knee flexion ≤ 90 degrees
* Pre-study clinical laboratory findings within the normal range or, if outside the normal range, deemed not clinically significant by the Investigator
* Able to swallow an oral suspension and in the opinion of the Investigator, is expected to continue to be able to do so for the duration of the trial. Administration via a feeding tube is not allowed.
* Forced vital capacity (FVC) > 20% predicted
* Male patients who have reached puberty must agree to do either of the following from Screening until 10 weeks after the last dose of the investigational product unless they have had a vasectomy and confirmed sperm count is zero:

  * Abstain from sexual intercourse, OR
  * If having heterosexual intercourse, must use a condom and their female partners who are of childbearing potential must use a highly effective contraception method*
* Female patients who have had their first period will be considered of childbearing potential unless they are anatomically and physiologically incapable of becoming pregnant. If of childbearing potential, the female patients must:

  * Have a negative urine/serum pregnancy test at Screening AND
  * Abstain from heterosexual intercourse from Screening until 10 weeks after the last dose of investigational product OR
  * If having heterosexual intercourse, must use a highly effective contraception method* and require the male partners to use a condom from Screening until 10 weeks after the last dose of investigational product

    *Highly effective contraception methods include:
  * Established use of oral, injected or implanted hormonal methods of contraception
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
* Male patients must agree to refrain from sperm donation from Screening until 10 weeks after the final study drug administration

Exclusion Criteria:

* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator
* Hospitalization within 2 months of Screening
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (appendectomy, hernia repair, and/or cholecystectomy will be allowed)
* A clinically significant illness within 4 weeks of Screening
* History of alcoholism or drug addiction within 2 years prior to Screening
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to Screening
* Patient has used a strong CYP3A4 inhibitor within 7 days prior to first dose of study drug or a strong CYP3A4 inducer within 14 days prior to first dose of study drug
* Any other medical condition that would interfere with performance of testing including (but not limited to) significant joint pain or arthritis limiting mobility, and chronic neuromuscular pain sufficient to require ongoing analgesic medication
* Participation by two people at the same time that are living in the same household
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days or five half-lives of the other investigational study drug, whichever is greater, prior to Screening
* An ALT or AST greater than 2-fold the upper limit of normal (ULN) or has total bilirubin greater than the ULN at screening. These assessments may be repeated once at the investigator's discretion (within the screening window)
* Currently taking nusinersen, or has taken it in the past, or plans to take it during the course the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Cytokinetics, Study Director — Cytokinetics, Inc.
Locations (19):
- United States (15):
  - UCLA, Los Angeles, California
  - University of California Irvine, Orange, California
  - Pediatric Neuromuscular Clinic Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - Nemours Childrens Hospital, Orlando, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hospital Institute for Clinical and Translational Research Pediatric Clinical Research Unit, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Utah, Clinical Neurosciences Center, Salt Lake City, Utah
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Children's Hospital - LHSC, London, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with SMA were enrolled at 18 sites in Canada and the United States. The first patient was enrolled on 14 January 2016 and the last patient completed on 31 May 2018.
Pre-assignment Details: Eligible patients were male or female, ≥12 y of age and had a genetically confirmed diagnosis of SMA. Ambulatory patients were able to walk ≥50 m in 6 min; and non-ambulatory patients were able to tolerate upright sitting with support for 3 h. Patients had an FVC >20% predicted, an HFMS-E score ≥10 and ≤54, and elbow and knee flexion ≤90 degrees.
Groups:
- Placebo: Patients randomized to this treatment arm received a placebo suspension twice daily for 8 weeks.
  Placebo: Granules for oral suspension (placebo)
- Reldesemtiv 150 mg Twice Daily: Patient randomized to this treatment arm received reldesemtiv suspension at a dose of 150 mg, twice daily for 8 weeks.
  Reldesemtiv 150 mg: Granules for oral suspension, 18.7% reldesemtiv
- Reldesemtiv 450 mg Twice Daily: Patients randomized to this treatment arm received reldesemtiv suspension at a dose of 450 mg, twice daily for 8 weeks.
  Reldesemtiv 450 mg: Granules for oral suspension, 56.0% reldesemtiv
Period: Overall Study
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Started | 26 | 24 | 20
Completed | 24 | 24 | 17
Not Completed | 2 | 0 | 3
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients randomized to this treatment arm received a placebo suspension twice daily for 8 weeks.
- Reldesemtiv 150 mg Twice Daily: Patient randomized to this treatment arm received reldesemtiv suspension at a dose of 150 mg, twice daily for 8 weeks.
- Reldesemtiv 450 mg Twice Daily: Patients randomized to this treatment arm received reldesemtiv suspension at a dose of 450 mg, twice daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily | Total
Number analyzed (Participants) | 26 | 24 | 20 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (16.03) | 27.8 (11.96) | 32.6 (17.92) | 29.4 (15.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 8 | 29
  Male | 15 | 14 | 12 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 22 | 23 | 18 | 63
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Time since SMA symptom onset [Mean (Standard Deviation); unit: months] | 302.5 (170.11) | 246.8 (105.93) | 299.8 (174.32) | 282.6 (152.56)
Time since genetically confirmed diagnosis [Mean (Standard Deviation); unit: months] | 139.2 (75.09) | 138.8 (81.45) | 101.4 (82.27) | 128.2 (80.06)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Forced Vital Capacity (FVC)
Description: FVC was measured using a calibrated spirometer (in units of liters). Patients were instructed to take as deep an inspiration as possible followed by a maximum exhalation (blowing out all the air in their lungs).
Time Frame: baseline and 8 weeks
Population: The analysis population includes patients who received at least 1 dose of reldesemtiv and had results from the relevant outcome measure at Week 8.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 25 | 24 | 18
liters | -0.02 (0.042) | -0.03 (0.043) | -0.07 (0.050)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.9086, Mixed Models Analysis; Least squares mean difference = -0.01, 95% CI 2-sided [-0.13 to 0.11], Standard Error of Mean 0.060
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.4361, Mixed Models Analysis; Least squares mean difference = -0.05, 95% CI 2-sided [-0.18 to 0.08], Standard Error of Mean 0.065

2. Primary Outcome: Change From Baseline to Week 8 in Maximum Inspiratory Pressure (MIP)
Description: MIP was measured (in units of cm H20) using a calibrated spirometer with an inspiratory pressure valve attached. For the test, patients were asked to inhale as forcefully as possible, to their maximum pressure.
Time Frame: baseline and 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm H2O
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 25 | 24 | 18
cm H2O | -2.62 (3.317) | -5.56 (3.401) | -1.63 (3.901)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.5382, Mixed Models Analysis; Least squares mean difference = -2.94, 95% CI 2-sided [-12.43 to 6.55], Standard Error of Mean 4.749
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.8464, Mixed Models Analysis; Least squares mean difference = 0.99, 95% CI 2-sided [-9.19 to 11.18], Standard Error of Mean 5.099

3. Primary Outcome: Change From Baseline to Week 8 in Maximum Expiratory Pressure (MEP)
Description: MEP was measured (in units of cm H20) using a calibrated spirometer with an exspiratory pressure valve attached. For the test, patients were asked to maximally inhale then perform a forced exhalation with as forcefully as possible.
Time Frame: baseline and 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm H2O
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 25 | 24 | 18
cm H2O | -4.22 (3.843) | 7.47 (3.941) | 8.93 (4.517)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.0378, Mixed Models Analysis; Least squares mean difference = 11.69, 95% CI 2-sided [0.68 to 22.70], Standard Error of Mean 5.506
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.0298, Mixed Models Analysis; Least squares mean difference = 13.15, 95% CI 2-sided [1.33 to 24.97], Standard Error of Mean 5.913

4. Primary Outcome: Muscle Strength Mega-Score at Week 8
Description: Muscle strength of 3 muscle groups (elbow flexion, knee extension, and shoulder abduction) were measured bilaterally using a hand-held dynamometer. Muscle strength was measured twice for each body location; if the variability between the 2 measures was > 15%, a third measure was obtained.
  The maximum muscle strength of the 2 measurements was identified and transformed as a percent change from baseline using the equation: ([postbaseline value - baseline value] / baseline value) × 100.
  The mega-score was a composite score that averaged strength across the 3 muscle groups. It was calculated as the mean of the non-missing transformed muscle strength scores among the 3 muscle groups each measure bilaterally (totaling 6 body locations).
Time Frame: baseline and 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 25 | 24 | 18
percent change | 14.34 (5.298) | 9.76 (5.393) | -0.88 (6.247)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.5461, Mixed Models Analysis; Least squares mean difference = -4.59, 95% CI 2-sided [-19.69 to 10.52], Standard Error of Mean 7.560
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.0672, Mixed Models Analysis; Least squares mean difference = -15.23, 95% CI 2-sided [-31.56 to 1.11], Standard Error of Mean 8.175

5. Primary Outcome: Change From Baseline to Week 8 in the Hammersmith Functional Motor Scale-Expanded (HFMS-E)
Description: The HFMS-E evaluated the level of independent mobility and motor skills through assessment of 33 test-items, each scored from 0 (worse) to 2 (better). The total score was calculated as the sum of the scores among the 33 test items, and has a range from 0 to 66.
Time Frame: baseline and 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 25 | 22 | 18
score on a scale | 1.40 (0.637) | 1.02 (0.675) | 0.39 (0.748)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.6849, Mixed Models Analysis; Least squares mean difference = -0.38, 95% CI 2-sided [-2.23 to 1.48], Standard Error of Mean 0.928
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.3091, Mixed Models Analysis; Least squares mean difference = -1.00, 95% CI 2-sided [-2.96 to 0.95], Standard Error of Mean 0.980

6. Primary Outcome: Change From Baseline to Week 8 in Revised Upper Limb Module (RULM)
Description: The RULM assessed motor function in the upper limbs (specifically shoulder, elbow, wrist, and hand function) that related to activities of everyday life. The RULM consisted of 20 items, 1 of which was scored on a 7-point scale (from 0 to 6), 18 were scored on a 3-point scale (from 0 to 2), and 1 was scored on a 2-point scale (0 or 1). The total score was the sum of each response and could range from a minimum of 0 to a maximum of 43 points. Higher scores reflected better motor function.
Time Frame: baseline and 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 25 | 24 | 18
score on a scale | 0.54 (0.397) | 1.15 (0.406) | 0.43 (0.468)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.2878, Mixed Models Analysis; Least squares mean difference = 0.61, 95% CI 2-sided [-0.53 to 1.75], Standard Error of Mean 0.571
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.8512, Mixed Models Analysis; Least squares mean difference = -0.12, 95% CI 2-sided [-1.34 to 1.11], Standard Error of Mean 0.616

7. Primary Outcome: Change From Baseline to Week 8 in the TUG Test
Description: The TUG test measured the time (in seconds) it took for a patient to rise from a chair, walk 3 meters, turn around, walk back to the chair and sit down.
Time Frame: baseline and 8 weeks
Population: This test was evaluated in ambulatory patients only.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 8 | 10 | 4
seconds | 0.24 (1.837) | -0.54 (1.708) | -2.87 (2.675)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.7612, Mixed Models Analysis; Least squares mean difference = -0.78, 95% CI 2-sided [-6.08 to 4.52], Standard Error of Mean 2.528
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.3502, Mixed Models Analysis; Least squares mean difference = -3.10, 95% CI 2-sided [-9.91 to 3.70], Standard Error of Mean 3.231

8. Primary Outcome: Change From Baseline to Week 8 in the 6MWT
Description: The 6MWT measured the distance (in meters) a patient walked in 6 minutes.
Time Frame: baseline and 8 weeks
Population: This test was evaluated in ambulatory patients only.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 9 | 12 | 6
meters | 1.39 (7.692) | 9.11 (6.826) | 26.28 (9.641)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.4684, Mixed Models Analysis; Least squares mean difference = 7.72, 95% CI 2-sided [-13.86 to 29.30], Standard Error of Mean 10.484
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.0584, Mixed Models Analysis; Least squares mean difference = 24.89, 95% CI 2-sided [-0.95 to 50.74], Standard Error of Mean 12.550

9. Primary Outcome: Patient Global Assessment at the End of Week 8
Description: Patients assessed whether they felt the same, better, or worse than prior to dosing on Day 1.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 25 | 24 | 18
Participants
  Better than pre-dose | 12 | 7 | 7
  Same as pre-dose | 13 | 15 | 11
  Worse than pre-dose | 0 | 2 | 0
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Odds ratio of active vs placebo comparison of the patients' global assessment of better than pre-dose vs same or worse than pre-dose; Test type: Superiority; p = 0.1686, Regression, Logistic; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.13 to 1.43]
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.5259, Regression, Logistic; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.20 to 2.30]

10. Primary Outcome: Investigator Global Assessment at the End of Week 8
Description: The Investigator assessed whether patient appeared the same, better, or worse than prior to dosing on Day 1.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 24 | 24 | 17
Participants
  Better than pre-dose | 6 | 7 | 6
  Same as pre-dose | 18 | 17 | 11
  Worse than pre-dose | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.7655, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.34 to 4.40]
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.4920, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.41 to 6.25]

11. Secondary Outcome: Reldesemtiv Maximum Observed Plasma Concentration (Cmax)
Description: Determined by evaluation of reldesemtiv plasma concentrations from blood samples collected prior to dosing and at 1, 3, and 6 hours following dosing
Time Frame: End of Week 8
Population: The analysis population includes all patients who had an evaluable reldesemtiv Cmax value at Week 8.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 23 | 15
microgram/milliliter | 1.40 (43.18) | 3.34 (48.77)

12. Secondary Outcome: Reldesemtiv Area Under the Plasma Concentration-time Curve From 0 to 12 Hours (AUC0-12)
Description: as for outcome 11
Time Frame: End of Week 8
Population: The analysis population includes patients who had an evaluable reldesemtiv AUC0-12 value at Week 8.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour x microgram/milliliter
Arm/Group | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Number analyzed (Participants) | 23 | 15
hour x microgram/milliliter | 9.0 (49.38) | 25.0 (52.19)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected over approximately 12 weeks: from administration of the first dose of study drug through the treatment period [8 weeks] and through the follow-up period [4 weeks after the last dose of study drug]).
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/24 | 2/20
Other Adverse Events (participants affected / at risk) | 24/26 | 20/24 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Reldesemtiv 150 mg Twice Daily (N=24) | Reldesemtiv 450 mg Twice Daily (N=20)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | Reldesemtiv 150 mg Twice Daily (N=24) | Reldesemtiv 450 mg Twice Daily (N=20)
Headache (Nervous system disorders) | 5 (5) | 6 (6) | 5 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (5) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 1 (2) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cystatin C increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bruxism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT02644668/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT02644668/SAP_001.pdf